CLINICAL TRIAL: NCT04392869
Title: Testing the Effects of Two Mindfulness-based Programs on Well Being and Academic Performance of Undergraduate Students of Translation and Interpreting: An Interventional Study
Brief Title: The Effects of Mindfulness-based Training in Undergraduate Students of Translation and Interpreting
Acronym: CRAFTftiugr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Chair in Conscience and Development (UGR) (Unknown); Mind, Brain and Behaviour Research Centre (CIMCYC) (Unknown)
Responsible Party: Principal Investigator, Mercedes García de Quesada, Mercedes García de Quesada, PhD Associate Professor-tenured, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PIBPD 431 (PPFID 2018-2020)
Record Dates: First submitted 2020-05-09; First posted 2020-05-19 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Psychological Distress; Life Stress; Anxiety; Perfectionism; Emotional Intelligence; Creativity; Attention; Empathy
Keywords: Academic Performance; Mindfulness; Learning in Higher Education; Emotional Regulation; Curriculum Design; Cognitive Behavioral Training; Translation and Interpreting Studies
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Emotional Regulation | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Students are randomly assigned to two groups: the MBSR group that receives an extended and adapted version of the MBSR program and the CRAFT group that receives an extended and adapted version of the CRAFT. All participants are asked to fill in an informed consent and a demographic questionnaire to determine eligibility. Eligible participants are randomly assigned to either the MBSR group or the CRAFT group. Both programs are taught simultaneously. The outcome measures will be evaluated against a third group who receives no intervention at all and could not be randomly assigned. This passive control group is formed with students from the same courses as experimental participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator: researchers have no information on participants' allocation in the groups; a research assistant from the Cognitive Neuroscience Group is designated for this purpose. None of the participants are students of any of the researchers. For the purpose of communicating with the participants over group allocation, another lecturer from the Translation Department is appointed. Outcome Assessors: all measures except one are collected online via the UGR LimeSurvey platform and no recording of group assignment is introduced in the system. The only face-to-face measure is administered at the baseline by another member who is blind to hypothesis. Care providers: they are not informed about the outcome measures or specific research hypothesis regarding expected effects for each program. Participants: although it is not possible to blind their assignment to the groups, they are not informed about the specific hypothesis regarding the expected outcomes of the programs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CRAFT group (Experimental): This arm will instruct the students on an adapted and extended version of the CRAFT program. This is a mindfulness based program which is a systematic combination of practices derived from ancient philosophies, such as yoga and Buddhism, in conjunction with more recent disciplines such as mindfulness, emotional intelligence and positive psychology. The contents are structured along in five consecutive modules aimed at cultivating and enhancing consciousness, relaxation and regulation, attention, bliss and transcendence.
  Interventions: Behavioral: The CRAFT program (adapted due to COVID-19)
- MBSR group (Experimental): This arm will instruct the students on an adapted and extended version of the Mindfulness-Based Stress Reduction (MBSR) program. The MBSR is a secular, evidence-based practice originally developed for chronic pain, but which has reported positive results among an array of clinical and nonclinical populations. This program aims to cultivate non-judgmental attention to and awareness of present moment experience while promoting stress reduction.
  Interventions: Behavioral: The MBSR program (adapted due to COVID-19)
- No intervention group (No Intervention): This group does not receive any instruction. The aim of this arm is to determine if there are any differences in outcomes between the two groups that receive intervention and this one.

INTERVENTIONS:
Behavioral: The CRAFT program (adapted due to COVID-19) — The CRAFT program was created by P. Posadas, PhD (Posadas 2017). This program aims to cultivate positive emotions toward oneself and others, engaging socio-emotional processes and activating traits such as empathy, motivation and creativity. It has been previously implemented in other Higher Education Institutions (Rull et al 2019, Posadas 2018, 2019).
  It originally consists of 8 weekly classes, 2 hours each (18 hours direct instruction) but it has been adapted and extended due to the situation caused by the COVID19 pandemic.
  The resulting 12 week program is structured along the following topics: Consciousness, Relaxation-Breathing-Regulation, Mindfulness/Full Attention, Bliss, Transcendence, Communication as Connection, Mindfully, Consciously and Blissfully Living our Daily Lives, My Work of Art "My Wonderful Craft Work Here and Now", Time and Energy Management, Passion and Compassion in the COVID context.
  Other Names: The CRAFT (Conscience, Relaxation-regulation, Attention, Bliss and Transcendence) program, adapted due to COVID-19
  Arms: CRAFT group
Behavioral: The MBSR program (adapted due to COVID-19) — The MBSR program is a group-based therapy which teaches mindfulness skills through a range of formal and informal mindfulness practices. Created by Kabat-Zinn (1982), in the current study it is taught by an officially accredited instructor and is compliant with the guidelines established by Brown University and the University of Massachusetts, USA.
  It originally consists of 8 weekly classes, 2 hours each (18 hours direct instruction) but it has been adapted and extended due to the situation caused by the COVID19 pandemic.
  The resulting 12 week program is structured along the following topics: The Underpinnings of MBSR, The Perception of Reality, Emotion Regulation, Understanding Stress: The Mind-Body Relation, Responding to Stress, Communication and Personal Relations, Daily Life Management, My Personal Plan: "The First Week of the Rest of my Life", Time and Energy Management, Emotion Regulation in the COVID context.
  Other Names: The MBSR (Mindfulness Based Stress Reduction) program, adapted due to COVID-19
  Arms: MBSR group

SUMMARY:
The Faculty of Translation and Interpreting of the University of Granada (UGR) has been leading the lists of the best faculties in this area in Spain and abroad for years. This has largely defined the profile of its students as high performing and, therefore, more prone to display maladaptive perfectionism which can lead to psychological distress (Rice et al 2006). However psychological distress is not something that only affects high profile students. Several studies report overall greater stress levels among undergraduate students when compared to general population levels (Ramasubramanian 2017). In fact, it is estimated that nearly 40 percent of university students experience mild to severe depressive symptoms with over 50 percent of students predicted to experience some level of depressive symptomatology during their college years (Pogrebtsova et al 2018: 46). Coping with cognitive and emotional challenges is therefore a desirable aim for every student on a daily bases.

It is within this framework that CRAFTftiugr was born, a teaching innovation project, which is the result of the interaction among experts in mindfulness, lecturers and researchers in Translation and Interpreting and Experimental Psychology, students, Administrative and Support Staff and social stakeholders in the context of Higher Education. The main objective of the study is to test whether participating in a course on mindfulness-based techniques can improve students' cognitive, emotional and personal traits as well as academic performance. Together with this main purpose, the present study also aims to compare the effects of two mindfulness based programs, MBSR and CRAFT, on the students' ability to improve specific aspects of cognition, emotional intelligence, creativity or academic performance among others. Both mindfulness-based programs involve training sustained attention and an accepting and open attitude though they differ in several aspects of their methods, intention and aims.

Drawing conclusions from the outcomes, a curriculum applied to Translation and Interpreting Studies will be designed aimed at preventing the development of psychological stress, perfectionism and other anxiety disorders, maximizing comfort in the Higher Education context and, ultimately, improving academic achievement.

DETAILED DESCRIPTION:
The first year of the project has been devoted to the design of the study, the creation of the curriculum content for the courses (see attached document), all the administrative procedures aimed at formally introducing a course of this type into the Bachelor's Degree in Translation and Interpreting, and applying and receiving approval from the UGR Ethics Committee on Human Research (CEIH), the UGR Human Subjects Protection Review Board (see attached document).

All 1st and 4th year students are informed and invited to participate both in the course and in the study; they can choose to participate either in the study alone, in the course alone or in both.

So that the 4 ECTS credits of the mindfulness-based course can be validated for the completion of the Degree in Translation and Interpreting as prescribed by the European Higher Education Area, a petition was filed to the governing body of the Faculty of Translation and Interpreting of the UGR. In this petition, the content of the course, design and aim of the study, potential participants, duration and other issues related with the project were included and explained. The Faculty grants some facilities (lecture rooms and Administrative and Support Staff's help) and allows the validation of 4 ECTS credits in exchange for participation in the course.

In order to encourage participation in the study besides the 4 European Credit Transfer and Accumulation System (ECTS) credits obtained as a result of attending the course, they could receive a discount on the original price for the ECTS credit in case they also opt for participating in the study. If they are grant holders, they get a further discount.

All participants are asked to fill in an informed consent, a demographic questionnaire to determine eligibility and a battery of tests. Eligible participants are randomly assigned to either the MBSR group or the CRAFT group. To ensure a balanced proportion of 1st and 4th year students in each group, the course year variable is blocked. Also, excluded students who follow the course, are assigned to both groups proportionally with the criterion of "being 1st or 4th year students".

All questionnaires are uploaded to the UGR LimeSuvey platform, an open source online survey tool specially designed to develop, publish and collect survey responses. This software is the one recommended by the University of Granada to present and collect online data for research purposes as it complies with all current legislation and ensures that all protection data requirements are being effectively met.

For specific security guarantees, an institutional email account is created through which all communication related to the project is carried out. In the same line, all the documentation generated within the project is uploaded and shared on a virtual cloud owned by the UGR (www.ugrdrive.ugr.es).

Both program instructors are fully qualified. Carmen Verdejo-Lucas (MA) is a certified MBSR instructor with more than 30 year experience. She is a clinical psychologist specialized in mindfulness and compassion based interventions. She is also a certified Cultivating Emotional Balance (CEB) instructor by Santa Barbara Institute for Consciousness Studies and has received training from some of the most outstanding figures in mindfulness and compassion: Jon Kabat-Zinn, Alan Wallace, Eve Eckman, Ronald Siegel, Paul Gilbert, Jonh Picock, Margaret Cullen and Gonzalo Brito. Pilar Posadas de Julián (PhD) is specialized in mindfulness in educational contexts. She did her degree in Translation and Interpreting, and her PhD in Linguistics and Language Learning. As a musician, she works as a full professor at the Department of Pedagogy and Singing of the Conservatoire for Music and Dance combining this job with university postgraduate lecturing at different universities and institutions in and outside Spain. With more than 30 year experience in yoga, meditation and relaxation techniques, she is an accredited practitioner in a variety of mindfulness and yoga based techniques. She has been IP in several teaching innovation projects and has been awarded different prizes.

Due to the health emergency crisis caused by the COVID-19 pandemic, following instructions by our university (https://covid19.ugr.es/), the original study design has been changed from crossover to parallel. Contents of the programs and teaching methodology have also changed accordingly to adapt to online classes. Both programs are adapted and extended due to the circumstances.

Data collection is done at two different points in time: 1, before initiating the intervention, and 2, at the end of the intervention. Both data gathering phases lasts for approximately 15 days.

At the baseline, the only face-to-face measure is administered as such by another member who is blind to hypothesis. Due to the exigencies of health emergency situation and the impossibility to administer this measure face to face at the end of the intervention, it is also uploaded to the LimeSurvey platform and administered online at the end of the intervention.

The University of Granada General Foundation was the entity appointed to carry out all the administrative procedures (participants' enrollment, payment of fees, participants' medical insurance, certificate issuing at the end of the course and the like). The Chair in Conscience and Development of the University of Granada (Spain) is responsible of co-funding and the study members from the Cognitive Neuroscience Group (HUM-379, https://www.ugr.es/~jcarlosresina/Home.html) at the Mind, Brain and Behavior Research Centre (CIMCYC) of the University of Granada (Spain) are responsible of randomization and data analysis.

It is expected to find improvements in all measures (psychological and academic) in both groups after completing the course compared to pre-training and compared to a passive control group (students from the same degree that didn't chose to receive the course during the present academic year). In order to measure potential specific effects of each mindfulness program, pre-training to post-training psychological measures will be compared once completed the first program. Altogether, this applied study might help to elucidate whether these important transversal competences and soft skills in Translation and Interpreting can improve with mindfulness-based techniques and ultimately could be recommended as part of the official curricula of the Translating and Interpreting degree.

ELIGIBILITY:
Inclusion Criteria:

* Students from 1st year of the joint Bachelor's Degree in Translation and Interpreting, and Tourism of the University of Granada.
* Students from 1st year of the Bachelor's Degree in Translation and Interpreting of the University of Granada.
* Students from 4th year of the Bachelor's Degree in Translation and Interpreting of the University of Granada.

Exclusion Criteria:

* Current psychotherapy or history of psychotic disorder or neurological condition.
* Established formal meditation prior experience.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change on the Five Facets Mindfulness Questionnaire | Baseline, 4 months
  A 39-item self-report scale, translated and validated in Spanish, that measures mindfulness traits (Baer et al 2006, 2010; Cebolla et al 2012). Respondents rate a series of statements on a 5-point likert scale, with 1 being "never" and 5 being "very often".
Change on the Emotion Regulation Questionnaire | Baseline, 4 months
  A 10-item self-report scale, translated and validated in Spanish, that measures emotion regulation (Gross and John 2003; Cabello, Salguero, Fernández-Berrocal and Gross 2013). Respondents rate a series of statements on a 7-point likert scale, with 1 being "I strongly disagree" and 7 being "I totally agree".
Change on the Depression Anxiety Stress Scale | Baseline, 4 months
  A 21-item self-report scale, translated and validated in Spanish, that measures depression, anxiety and stress levels (Henry and Crawford 2005, Bados et al. 2005). Respondents rate a series of statements on a 4-point likert scale, with 0 being "not at all true of me" and 3 being "very true of me".
Change on the Trait Emotional Intelligence Questionnaire | Baseline, 4 months
  A 30-item self-report scale, translated and validated in Spanish, that measures self-regulation, psychological wellbeing, sociability and emotionality (Petrides et al 2016, Pérez 2003). Respondents rate a series of statements on a 7-point likert scale, with 1 being "I strongly disagree" and 7 being "I totally agree".
Change on the Cultural Intelligence Scale | Baseline, 4 months
  A 20-item self-report scale, translated and validated in Spanish, that measures cultural intelligence (Ang et al 2007; Moyano et al 2014). Respondents rate a series of statements on a 7-point likert scale, with 1 being "I strongly disagree" and 7 being "I totally agree".
Change on the Mind Wandering questionnaire | Baseline, 4 months
  An 8-item self-report scale, translated and validated in Spanish, that measures the levels of the mind wandering trait (Carriere et al 2013). Respondents rate a series of statements on a 7-point likert scale, with 1 being "almost never" and 7 being "almost always".
Change on the ANTIVEA task | Baseline, 4 months
  Online cognitive test, assessing several objective indices (based on participant's reaction times and accuracy) of attention and vigilance (Luna et al 2018).
Change on the Test on creativity | Baseline, 4 months
  Face-to-face questionnaire, in Spanish, measuring divergent thinking (Berná and Limiñana 2010, Elisondo et al 2017).
Change on the Motivated Strategies for Learning Questionnaire | Baseline, 4 months
  A 52-item self-report scale, translated and validated in Spanish, that measures motivation and learning strategies (Rojas-Ospina and Valencia-Serrano 2019; Muñoz and Asencio 2018; Pintrich et al 1987, Pintrich and De Groot 1990; Martínez Fernández and Galán 2000). Respondents rate a series of statements on a 5-point likert scale, with 1 being "I strongly disagree" and 5 being "I totally agree".

SECONDARY OUTCOMES:
Academic performance assessment | Up to 4 years
  Results from primary outcome are associated with academic performance of students' core subjects.
Qualitative questionnaire on students' experience | 4 months
  This qualitative questionnaire with open ended questions builds directly on the results from the quantitative phase. The quantitative results are interpreted in more detail through the qualitative data.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Translation and Interpreting of the University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data set from the ANTI-VEA task (one of our primary outcomes) will become part of a more general database belonging to the UGR Cognitive Neuroscience research group (HUM-379). This group is responsible for the design of the task with the aim to study attentional processes. Three of the researchers from the present project belong to such research team.
Time Frame: From data collection.
Access Criteria: Data set from the ANTI-VEA task will only be shared anonymized.

REFERENCES:
- [Background] Baer RA, Samuel DB, Lykins EL. Differential item functioning on the Five Facet Mindfulness Questionnaire is minimal in demographically matched meditators and nonmeditators. Assessment. 2011 Mar;18(1):3-10. doi: 10.1177/1073191110392498. Epub 2010 Dec 30. PMID 21193491
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Carriere JSA, Seli P, Smilek D. Wandering in both mind and body: individual differences in mind wandering and inattention predict fidgeting. Can J Exp Psychol. 2013 Mar;67(1):19-31. doi: 10.1037/a0031438. PMID 23458548
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Luna FG, Marino J, Roca J, Lupianez J. Executive and arousal vigilance decrement in the context of the attentional networks: The ANTI-Vea task. J Neurosci Methods. 2018 Aug 1;306:77-87. doi: 10.1016/j.jneumeth.2018.05.011. Epub 2018 May 20. PMID 29791865
- [Background] Pogrebtsova E, Craig J, Chris A, O'Shea D, Gonzalez-Morales MG. Exploring daily affective changes in university students with a mindful positive reappraisal intervention: A daily diary randomized controlled trial. Stress Health. 2018 Feb;34(1):46-58. doi: 10.1002/smi.2759. Epub 2017 May 17. PMID 28512859
- [Background] Ang S, Van Dyne L, Koh C, Ng KY, Templer KJ, Tay C, Chandrasekar NA. Cultural intelligence: Its measurement and effects on cultural judgment and decision making, cultural adaptation and task performance. Manage Organ Rev [Internet]. 2007; 3(3): 335-71. Available from: www.scopus.com
- [Background] Berná JC, Limiñana Gras RM. The genie in a bottle. the CREA test, questions and creativity. introduction to special theme
- [Background] Cabello R, Salguero JM, Fernández-Berrocal P, Gross JJ. A Spanish adaptation of the emotion regulation questionnaire. Eur J Psychol Assess [Internet]. 2013; 29(4): 234-40. Available from: www.scopus.com
- [Background] Elisondo RC, Donolo DS, Limiñana-Gras RM. The measure of originality in CREA test responses. An Psicol [Internet]. 2018; 34(1): 197-210. Available from: www.scopus.com
- [Background] Martínez Fernández JR and Galán F. Estrategias de aprendizaje, motivación y rendimiento académico en alumnos universitarios. Revista Española de Orientación y Psicopedagogía. 2000; 11(19): 35-50.
- [Background] Moyano M, Tabernero C, Melero R, Trujillo HM. Spanish version of the cultural intelligence scale (CQS). Rev Psicol Soc [Internet]. 2014; 30(1): 182-216. Available from: www.scopus.com
- [Background] Muñoz GN, Asencio EN. Improvement of self-regulation learning strategies at university: The impact of a program of academic fit to the degree. Bordon, Rev Pedagog [Internet]. 2018; 70(4): 121-36. Available from: www.scopus.com
- [Background] Petrides KV, Mikolajczak M, Mavroveli S, Sanchez-Ruiz M-, Furnham A, Pérez-González J-. Developments in trait emotional intelligence research. Emot Rev [Internet]. 2016; 8(4): 335-41. Available from: www.scopus.com
- [Background] Pintrich PR, De Groot EV. Motivational and self-regulated learning components of classroom academic performance. J Educ Psychol [Internet]. 1990; 82(1): 33-40. Available from: www.scopus.com
- [Background] Pintrich PR, McKeachie WJ, Smith DAF, Doljanac R, Lin YG, Naveh-Benjamin M, Crooks T, Karabenick S. The Motivated strategies for learning questionnaire. Ann Arbor, MI: University of Michigan, National Center for Research to Improve Postsecondary Teaching and Learning (NCRIPTAL); 1987.
- [Background] Posadas P. Mindfulness para músicos. Programa CRAFT. In: Lag López N, editor. Educación Musical: Recursos para el cambio metodológico. Málaga: Procompal Publicaciones; 2018. p. 221-226.
- [Background] Posadas P, inventor. Programa CRAFT en el marco del Proyecto MACF (Mundo Atento Consciente y Feliz) basado en Mindfulness, Yoga, Psicología Positiva y Sugestopedia orientado a las Enseñanzas de Régimen Especial: Enseñanzas Artísticas e Idiomas.
- [Background] Posadas P. Programa CRAFT. Mindfulness, Inteligencia Emocional, Psicología Positiva y Yoga en Educación. Granada: Educatori; 2019.
- [Background] Ramasubramanian S. Mindfulness, stress coping and everyday resilience among emerging youth in a university setting: A mixed methods approach. Int J Adolesc Youth [Internet]. 2017; 22(3): 308-21. Available from: www.scopus.com
- [Background] Rice KG, Leever BA, Christopher J, Porter JD. Perfectionism, stress, and social (dis)connection: A short-term study of hopelessness, depression, and academic adjustment among honors students. J Couns Psychol [Internet]. 2006; 53(4): 524-34. Available from: www.scopus.com
- [Background] Rojas-Ospina T, Valencia-Serrano M. Adaptation and validation of a questionnaire on motivation self-regulation strategies in college students. Psykhe [Internet]. 2019; 28(1): 1-15. Available from: www.scopus.com
- [Background] Rull LM, de Julián MPP, Martín JLO. Learn English to the rhythm of Bach: An eclectic methodology for learning English based on suggestopedia and the CRAFT program. Int J Pedagogy Curric [Internet]. 2019; 26(1): 1-15. Available from: www.scopus.com
- [Background] Pérez JC. Adaptación y validación española del "Trait Emotional Intelligence Questionnaire"(TEIQue) en población universitaria. Encuentros en Psicología Social. 2003; 1(5): 278-283.
- [Result] Cásedas L, Funes MJ, Ouellet M, García de Quesada M. Training transversal competences in a bachelor's degree in translation and interpreting: preliminary evidence from a clinical trial. The Interpreter and Translator Trainer. 2022. DOI: 0.1080/1750399X.2022.2148964
- See also: Limesurvey open source survey tool — http://www.limesurvey.org
- Available data/document: Summary and comparison of mindfulness based programs: clinicaltrialsCRAFT — https://drive.ugr.es/index.php/s/ytdazx47iReHMeu — This is not a comprehensive description of any of the programs, but rather a schematic outline with the most salient similarities and differences between them.
- Available data/document: Human Subjects Review: clinicaltrialsCRAFT — https://drive.ugr.es/index.php/s/DGKxnBhZfm058DA — Human Subjects Review approval and its translation into English
- Available data/document: Informed Consent Form: clinicaltrialsCRAFT — https://drive.ugr.es/index.php/s/10ptY8LrAdwdWTj — This document contains the welcome email, the informed consent form and the demographic survey. Please, bear in mind that this is the English version of the text in Spanish uploaded to the LimeSurvey platform.
- Available data/document: Official CRAFTftiugr logo: clinicaltrialsCRAFT — https://drive.ugr.es/index.php/s/zHklhje0InjZAF7 — This is the official logo of the project. It represents a way of communication that goes beyond words. Earphones are a special reference to interpreters.